CLINICAL TRIAL: NCT06542692
Title: Effect of Whole Body Vibration Therapy on Pain, Muscle Strength, Balance and Quality of Life in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burak Çetinkaya (Other)
Responsible Party: Sponsor-Investigator, Burak Çetinkaya, principal investigator, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E68869993-511.06.01.01-1193507
Record Dates: First submitted 2024-07-19; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis
Keywords: vibration; whole body vibration; Osteoarthritis; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Whole body vibration therapy added group
  Interventions: Device: Whole Body Vibration; Device: physical therapy modalities
- control group (Experimental)
  Interventions: Device: physical therapy modalities

INTERVENTIONS:
Device: Whole Body Vibration — treatment duration, frequency
  Other Names: physical therapy modalities
  Arms: study group
Device: physical therapy modalities — ultrasound, hot pack, tens

SUMMARY:
The aim of this study is to examine the effects of whole body vibration therapy on knee osteoarthritis. While the participants did static exercise in one group, whole body vibration therapy was applied during static exercise in another group. As a result of 15 sessions of treatment in both groups, the effects on pain, muscle strength, balance and quality of life were compared.

ELIGIBILITY:
Inclusion Criteria:

* Those who were diagnosed with primary symptomatic knee OA according to ACR criteria,Ages between 35 and 70, Body mass index (BMI) ⩽35, Grade II or III according to Kellgren & Lawrence scale, Patients with persistent symptoms such as pain and stiffness for at least 3 months were included.

Exclusion Criteria:

* Those who have had knee surgery before, Those with central nervous system disease (especially epilepsy and serious psychotic disorders), those with a history of acute arthritis, Those with a history of DVT in the last 24 weeks, Those with advanced lung or heart disease (COPD and heart failure), Those diagnosed with inflammatory rheumatic diseases (Rheumatoid arthritis, Spondyloarthropathy, etc.), Patients diagnosed with advanced stage cancer were excluded from the study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
visual analog scala | 3 weeks
  Scale ranging from 0 to 10 points, where 0 points indicate no pain and 10 points indicate maximum pain.
Womac | 3 weeks
  Western Ontario and McMaster Universities Osteoarthritis Index
muscle strength | 3 weeks
  isometric muscle strength measurement(knee extension, flexion)
Biodex | 3 weeks
  Balance test
Short Form 36 | 3 weeks
  A test consisting of 36 questions to assess quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No